CLINICAL TRIAL: NCT00081497
Title: Multi-Center, Open-Label Study of the Safety and Efficacy of Fabrazyme in Patients With Fabry Disease That Previously Participated in the AGAL-008-00 Study
Brief Title: A Study of the Safety and Efficacy of Fabrazyme in Patients With Fabry Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGAL02503
Record Dates: First submitted 2004-04-14; First posted 2004-04-16 (Estimated); Results first posted 2010-08-18 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Fabry Disease
Keywords: alpha-galactosidase A; a-GAL; r-haGAL; Fabry; GL-3; Fabrazyme
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

ARMS (1):
- Fabrazyme 1.0 mg/kg every 2 weeks (Experimental): This is an open-label extension study to AGAL-008-00 (NCT00074984) and all patients received Fabrazyme treatment.
  Interventions: Biological: agalsidase beta

INTERVENTIONS:
Biological: agalsidase beta — 1.0 mg/kg every 2 weeks
  Other Names: Fabrazyme; r-hαGAL

SUMMARY:
People with Fabry Disease have an alteration in their genetic material (DNA) which causes a deficiency of the alpha-galactosidase A enzyme. Fabrazyme (agalsidase beta) is a drug that helps to break down and removes certain types of fatty substances called "glycolipids". These glycolipids are normally present within the body in most cells. In Fabry disease, glycolipids build up in various tissues such as the liver, kidney, skin, and blood vessels because a-galactosidase A is not present, or is present in small quantities. The build up of glycolipid (globatriaosylceramide or GL-3) levels in these tissues in particular is thought to cause the clinical symptoms that are common to Fabry disease. This study analyzed the safety and efficacy of Fabrazyme in the treatment of patients with Fabry disease that previously participated in the AGAL-008-00 (NCT0074984) study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have successfully completed the previous double-blind study AGAL-008-00 (NCT00074984)
* Patients must provide written informed consent prior to study participation
* Female patients of childbearing potential must have a negative pregnancy test prior to each dosing and all female patients must use a medically accepted form of contraception throughout the study

Exclusion Criteria:

* The patient was unable to complete AGAL-008-00 (NCT00074984)
* The patient has undergone kidney transplantation or is currently on dialysis
* The patient has diabetes mellitus or presence of confounding renal disease
* The patient has a clinically significant organic disease or an unstable condition that precludes participation
* The patient is unwilling to comply with the protocol requirements

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2004-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (25):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of San Francisco, San Francisco, California
  - University of Connecticut Health Partners, West Hartford, Connecticut
  - Oncology Hematology Association, Coral Springs, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Gene Therapy Center - Department of Pediatrics and Institute of Human Genetics, Minneapolis, Minnesota
  - Children's Hospital, Buffalo, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester School of Medicine, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Washington School of Medicine, Seattle, Washington
- Canada (3):
  - Queen Elizabeth II Health Center, Halifax, Nova Scotia
  - North York General Hospital, Toronto, Ontario
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
- University Hospital, Prague, Czechia
- Sopron Megyei Jogu Varos Erzsebet Korhaz, Sopron, Hungary
- Klinika Chorob Metabolicznych Instytut, Warsaw, Poland
- Hope Hospital, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only those patients who successfully completed the AGAL-008-00 (NCT00074984) trial were eligible for participation in the AGAL02503 (NCT00081497) extension study.
Groups:
- Placebo/Fabrazyme: Patients who had been randomized to placebo during AGAL-008-00 (NCT00074984) and were then transitioned to open-label Fabrazyme (1.0 mg/kg every 2 weeks) prior to or at entry to AGAL02503 (NCT00081497).
- Fabrazyme/Fabrazyme: Patients who had been randomized to Fabrazyme in AGAL-008-00 (NCT00074984) and were then transitioned to open-label Fabrazyme (1.0 mg/kg every 2 weeks) prior to or at entry into AGAL02503 (NCT00081497).
Period: Overall Study
Arm/Group | Placebo/Fabrazyme | Fabrazyme/Fabrazyme
Started | 28 (Patients who were randomized to placebo in AGAL-008-00 (NCT00074984).) | 39 (Patients who were randomized to Fabrazyme in AGAL-008-00 (NCT00074984).)
Completed | 25 | 37
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Fabrazyme | Fabrazyme/Fabrazyme | Total
Number analyzed (Participants) | 28 | 39 | 67
Age, Customized [Number; unit: participants]
  <40 years | 8 | 7 | 15
  ≥40 years | 20 | 32 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (9.31) | 46.6 (9.72) | 45.3 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 24 | 34 | 58
Race/Ethnicity [Number; unit: participants]
  Caucasian | 24 | 35 | 59
  Black | 0 | 0 | 0
  Hispanic | 2 | 3 | 5
  Asian | 1 | 1 | 2
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Difference in Inverse Serum Creatinine Within Patients' Slopes Between the Placebo AGAL-008-00 (NCT00074984) and Fabrazyme AGAL02503 (NCT00081497) Periods
Description: The primary efficacy analysis was the summary of change in slope of inverse serum creatinine for Placebo/Fabrazyme patients in the Intent to Treat (ITT) Population. It compared the placebo period slope with the Fabrazyme period slope.
Time Frame: Placebo period AGAL-008-00 (up to 35 months) through Fabrazyme period AGAL02503 (18 months)
Population: ITT Population - Analysis compares results during the placebo period with those during the Fabrazyme period and includes only the 28 patients who were randomized to placebo in the AGAL-008-00 (NCT00074984) study; as such no formal sample size calculations were performed.
Measure: Least Squares Mean (Standard Error); unit: dL/mg/year
Groups:
- Placebo Period - AGAL-008-00 (NCT00074984): Patients who had been randomized to placebo during AGAL-008-00 (NCT00074984).
- Fabrazyme Period - AGAL02503 (NCT00081497): Placebo patients who had been transitioned to open-label Fabrazyme prior to or at entry into AGAL02503 (NCT00081497). 1.0 mg/kg of Fabrazyme given to the patients every 2 weeks for 18 months.
Arm/Group | Placebo Period - AGAL-008-00 (NCT00074984) | Fabrazyme Period - AGAL02503 (NCT00081497)
Number analyzed (Participants) | 28 | 28
dL/mg/year | -0.044 (0.012) | -0.073 (0.011)
Statistical Analysis 1: Comparison: Placebo Period - AGAL-008-00 (NCT00074984) vs Fabrazyme Period - AGAL02503 (NCT00081497); The statistical analysis represents the primary outcome measure results; Test type: Superiority or Other; p = 0.0130, Mixed Models Analysis; Mixed effects model with a population level (fixed effect) intercept and slope and a subject level (random effect) intercept and slope; Change in Slope Mean = -0.029, 95% CI [-0.051 to -0.007]

2. Post Hoc Outcome: Differences in Slopes of Estimated Glomerular Filtration Rate (eGFR) Comparing Randomized Placebo vs Fabrazyme Patients (Based on the Original Randomization in AGAL-008-00 (NCT00074984)) by Baseline eGFR Subgroups of >60 and ≤60 mL/Min/1.73 m^2.
Description: Summary of differences in slopes of eGFR comparing randomized placebo vs Fabrazyme patients by baseline eGFR subgroups. Differences in slopes are the placebo slope minus the Fabrazyme slope. Therefore, a negative difference indicates a greater decline in the placebo patients relative to the Fabrazyme patients.
Time Frame: Throughout study; 18 months
Population: ITT population. For subgroup Estimated Glomerular Filtration Rate (eGFR) >60, there were 9 placebo patients and 15 Fabrazyme patients. For subgroup eGFR ≤60, there were 19 placebo patients and 24 Fabrazyme patients. For randomized Fabrazyme patients, both the double-blind and open-label data was used.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2/year
Groups:
- Placebo - AGAL-008-00 (NCT00074984) eGFR >60: Patients who had been randomized to placebo during AGAL-008-00 (NCT00074984) using only placebo period data from the AGAL-008-00 (NCT00074984) study.
- Fabrazyme - AGAL02503 (NCT00081497) eGFR >60; Fabrazyme - AGAL02503 (NCT00081497) eGFR ≤60: Patients who had been randomized to Fabrazyme in AGAL-008-00 (NCT00074984) and were then transitioned to open-label Fabrazyme prior to or at entry into AGAL02503 (NCT00081497) using all Fabrazyme treatment period data from the AGAL00800 (NCT00074984) and AGAL02503 (NCT00081497) studies.
- Placebo - AGAL-008-00 (NCT00074984) eGFR ≤60: Patients who had been randomized to placebo during AGAL-008-00 (NCT00074984) and were then transitioned to open-label Fabrazyme prior to or at entry to AGAL02503 (NCT00081497) using only placebo period data from the AGAL-008-00 (NCT00074984) study.
Arm/Group | Placebo - AGAL-008-00 (NCT00074984) eGFR >60 | Fabrazyme - AGAL02503 (NCT00081497) eGFR >60 | Placebo - AGAL-008-00 (NCT00074984) eGFR ≤60 | Fabrazyme - AGAL02503 (NCT00081497) eGFR ≤60
Number analyzed (Participants) | 9 | 15 | 19 | 24
mL/min/1.73m^2/year | -7.685 (1.836) | -0.898 (1.129) | -2.575 (1.188) | -4.906 (0.900)
Statistical Analysis 1: Comparison: Placebo - AGAL-008-00 (NCT00074984) eGFR >60 vs Fabrazyme - AGAL02503 (NCT00081497) eGFR >60; Statistical Analysis 1 represents the post-hoc outcome results for difference in slope mean of eGFR subgroup >60; Test type: Superiority or Other; p = 0.0027, Mixed Effects Model; Mean Difference = -6.787, 95% CI [-11.123 to -2.450]
Statistical Analysis 2: Comparison: Placebo - AGAL-008-00 (NCT00074984) eGFR ≤60 vs Fabrazyme - AGAL02503 (NCT00081497) eGFR ≤60; Statistical Analysis 2 represents the post-hoc outcome results for difference in slope mean of eGFR subgroup ≤ 60; Test type: Superiority or Other; p = 0.1268, Mixed Effects Model; Mean Difference = 2.330, 95% CI [-0.685 to 5.345]

3. Secondary Outcome: Serum Creatinine at Pre-Fabrazyme and 6, 12, and 18 Months
Description: Pre-Fabrazyme=baseline visit of AGAL-008-00 (NCT00074984) for Fabrazyme patients; assessment prior to open-label for placebo patients who transitioned to Fabrazyme in AGAL-008-00 (NCT00074984); assessment prior to first Fabrazyme infusion in AGAL02503 (NCT00081497) for placebo patients who did not transition to Fabrazyme in AGAL-008-00 (NCT00074984).
Time Frame: Pre-Fabrazyme, 6, 12, and 18 months
Population: ITT population-67 patients had assessments at 6 and 12 months while 65 patients had assessments at 18 months in the open-label extension study.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Fabrazyme 1.0 mg/kg Every 2 Weeks: 1.0 mg/kg of Fabrazyme given to the patients every 2 weeks for 18 months. This is an open-label extension study to AGAL-008-00 (NCT00074984) and all patients received Fabrazyme treatment.
Arm/Group | Fabrazyme 1.0 mg/kg Every 2 Weeks
Number analyzed (Participants) | 67
mg/dL
  Serum Creatinine at Pre-Fabrazyme | 1.7 (0.60)
  Serum Creatinine at 6 months post-treatment | 1.8 (0.77)
  Serum Creatinine at 12 months post-treatment | 1.9 (0.98)
  Serum Creatinine at 18 months post-treatment | 2.1 (1.21)

4. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) at Pre-Fabrazyme and 6, 12, and 18 Months
Description: Pre-Fabrazyme=baseline visit of AGAL-00-800 (NCT00074984) for Fabrazyme patients; assessment prior to open-label for placebo patients who transitioned to Fabrazyme in AGAL-008-00 (NCT00074984); assessment prior to first Fabrazyme infusion in AGAL02503 (NCT00081497) for placebo patients who did not transition to Fabrazyme in AGAL-008-00 (NCT00074984).
Time Frame: Pre-Fabrazyme, 6, 12, and 18 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ml/min/1.73m^2
Arm/Group | Fabrazyme 1.0 mg/kg Every 2 Weeks
Number analyzed (Participants) | 67
ml/min/1.73m^2
  eGFR at Pre-Fabrazyme | 53.1 (19.62)
  eGFR at 6 months post-treatment | 52.6 (23.24)
  eGFR at 12 months post-treatment | 50.4 (22.73)
  eGFR at 18 months post-treatment | 47.8 (23.62)

5. Secondary Outcome: Plasma Globotriaosylceramide (GL-3) (Normal Plasma GL-3 Level is ≤ 7.03 µg/mL) at Pre-Fabrazyme and 6, 12, and 18 Months
Description: Pre-Fabrazyme=baseline visit of AGAL00800 for Fabrazyme patients; assessment prior to open-label for placebo patients who transitioned to Fabrazyme in AGAL00800; assessment prior to first Fabrazyme infusion in AGAL02503 for placebo patients who did not transition to Fabrazyme in AGAL00800.
Time Frame: Pre-Fabrazyme and 6, 12, and 18 months
Population: ITT population-64 patients had assessments at 6 and 18 months while 65 patients had assessments at 12 months in the open-label extension study.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Fabrazyme 1.0 mg/kg Every 2 Weeks
Number analyzed (Participants) | 65
µg/mL
  Plasma GL-3 at Pre-Fabrazyme | 9.0 (3.35)
  Plasma GL-3 at 6 months post-treatment | 4.8 (1.76)
  Plasma GL-3 at 12 months post-treatment | 4.7 (1.59)
  Plasma GL-3 at 18 months post-treatment | 4.6 (1.82)

6. Secondary Outcome: Proteinuria at Pre-Fabrazyme and 6, 12, and 18 Months
Description: as for outcome 3
Time Frame: Pre-Fabrazyme and 6, 12, and 18 months
Population: ITT population-62 patients had assessments at 6 months, 61 patients had assessments at 12 months, and 54 patients had assessments at 18 months in the open-label extension study.
Measure: Mean (Standard Deviation); unit: urine protein(mg/dL) / creatinine(mg/dL)
Arm/Group | Fabrazyme 1.0 mg/kg Every 2 Weeks
Number analyzed (Participants) | 62
urine protein(mg/dL) / creatinine(mg/dL)
  Proteinuria at Pre-Fabrazyme | 1.3 (1.46)
  Proteinuria at 6 months post-treatment | 1.1 (1.19)
  Proteinuria at 12 months post-treatment | 1.3 (1.77)
  Proteinuria at 18 months post-treatment | 1.3 (1.55)

ADVERSE EVENTS:
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Fabrazyme/Fabrazyme | Placebo/Fabrazyme | Total
Serious Adverse Events (participants affected / at risk) | 19/39 | 12/28 | 31/67
Other Adverse Events (participants affected / at risk) | 39/39 | 27/28 | 66/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fabrazyme/Fabrazyme (N=39) | Placebo/Fabrazyme (N=28) | Total (N=67)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 2
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2
Chest pain (General disorders) | 3 | 1 | 4
Pyrexia (General disorders) | 2 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 3 | 0 | 3
Kidney transplant rejection (Immune system disorders) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1 | 1
Localised infection (Infections and infestations) | 1 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Streptococcal infection (Infections and infestations) | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 1
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 1
Skin test positive (Investigations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 2
Nephritis interstitial (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 1 | 2
Renal impairment (Renal and urinary disorders) | 1 | 1 | 2
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fabrazyme/Fabrazyme (N=39) | Placebo/Fabrazyme (N=28) | Total (N=67)
Anaemia (Blood and lymphatic system disorders) | 5 | 5 | 10
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 2
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocythaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 3
Atrial flutter (Cardiac disorders) | 0 | 1 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 0 | 2
Bundle branch block left (Cardiac disorders) | 1 | 0 | 1
Bundle branch block right (Cardiac disorders) | 4 | 0 | 4
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 2
Cardiomegaly (Cardiac disorders) | 1 | 0 | 1
Dilatation atrial (Cardiac disorders) | 1 | 1 | 2
Dilatation ventricular (Cardiac disorders) | 1 | 0 | 1
Heart valve insufficiency (Cardiac disorders) | 1 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 4 | 0 | 4
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 3 | 0 | 3
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 5 | 0 | 5
Ventricular dysfunction (Cardiac disorders) | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 1 | 2
Ventricular hypertrophy (Cardiac disorders) | 3 | 1 | 4
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Ventricular wall thickening (Cardiac disorders) | 2 | 0 | 2
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 | 0 | 1
Exomphalos (Congenital, familial and genetic disorders) | 0 | 1 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 2 | 3
Deafness (Ear and labyrinth disorders) | 1 | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 1
Ear canal erythema (Ear and labyrinth disorders) | 1 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 6 | 3 | 9
Hearing impaired (Ear and labyrinth disorders) | 3 | 0 | 3
Hypoacusis (Ear and labyrinth disorders) | 4 | 0 | 4
Otorrhoea (Ear and labyrinth disorders) | 1 | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 5 | 0 | 5
Vertigo (Ear and labyrinth disorders) | 4 | 2 | 6
Hyperparathyroidism (Endocrine disorders) | 1 | 1 | 2
Binocular eye movement disorder (Eye disorders) | 2 | 0 | 2
Blepharitis (Eye disorders) | 1 | 0 | 1
Blepharospasm (Eye disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 1
Chalazion (Eye disorders) | 1 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 2 | 2
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 1
Conjunctival oedema (Eye disorders) | 1 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 1
Eye discharge (Eye disorders) | 1 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 1
Eyelid oedema (Eye disorders) | 2 | 0 | 2
Lacrimation increased (Eye disorders) | 0 | 2 | 2
Ocular hyperaemia (Eye disorders) | 1 | 0 | 1
Ocular hypertension (Eye disorders) | 1 | 0 | 1
Retinopathy (Eye disorders) | 2 | 0 | 2
Scleral haemorrhage (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 1 | 3 | 4
Visual acuity reduced (Eye disorders) | 1 | 0 | 1
Visual disturbance (Eye disorders) | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 12 | 3 | 15
Abdominal pain lower (Gastrointestinal disorders) | 5 | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 4 | 5 | 9
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 1
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 1 | 4
Defaecation urgency (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 6 | 18
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 1 | 6
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 1
Faeces pale (Gastrointestinal disorders) | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 3 | 1 | 4
Gastric disorder (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 2
Gingival pain (Gastrointestinal disorders) | 2 | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 1
Lip blister (Gastrointestinal disorders) | 0 | 1 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 13 | 11 | 24
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 1
Oral soft tissue disorder (Gastrointestinal disorders) | 0 | 1 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 1 | 2
Retching (Gastrointestinal disorders) | 1 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 5 | 2 | 7
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 6 | 1 | 7
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 1
Uvulitis (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 13 | 13 | 26
Adverse event (General disorders) | 10 | 3 | 13
Asthenia (General disorders) | 4 | 4 | 8
Axillary pain (General disorders) | 1 | 0 | 1
Catheter site haematoma (General disorders) | 1 | 0 | 1
Catheter site related reaction (General disorders) | 1 | 0 | 1
Chest discomfort (General disorders) | 3 | 3 | 6
Chest pain (General disorders) | 5 | 4 | 9
Chills (General disorders) | 20 | 12 | 32
Cyst rupture (General disorders) | 1 | 0 | 1
Discomfort (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 14 | 4 | 18
Feeling cold (General disorders) | 5 | 4 | 9
Feeling hot (General disorders) | 1 | 0 | 1
Feeling hot and cold (General disorders) | 1 | 0 | 1
Feeling jittery (General disorders) | 0 | 1 | 1
Gait disturbance (General disorders) | 1 | 0 | 1
Influenza like illness (General disorders) | 3 | 0 | 3
Infusion site bruising (General disorders) | 0 | 1 | 1
Infusion site reaction (General disorders) | 0 | 1 | 1
Injection site thrombosis (General disorders) | 1 | 0 | 1
Malaise (General disorders) | 1 | 1 | 2
Oedema (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 16 | 12 | 28
Pain (General disorders) | 11 | 5 | 16
Pitting oedema (General disorders) | 3 | 0 | 3
Pyrexia (General disorders) | 17 | 10 | 27
Sensation of foreign body (General disorders) | 0 | 1 | 1
Suprapubic pain (General disorders) | 1 | 0 | 1
Thirst (General disorders) | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 2 | 1 | 3
Abscess oral (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 6 | 3 | 9
Bronchitis acute (Infections and infestations) | 1 | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1 | 1
Catheter site infection (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 2 | 1 | 3
Conjunctivitis infective (Infections and infestations) | 1 | 0 | 1
Dental caries (Infections and infestations) | 2 | 0 | 2
Ear infection (Infections and infestations) | 1 | 2 | 3
Fungal infection (Infections and infestations) | 5 | 0 | 5
Gastroenteritis (Infections and infestations) | 2 | 1 | 3
Gastroenteritis viral (Infections and infestations) | 2 | 1 | 3
Gingival infection (Infections and infestations) | 2 | 0 | 2
Herpes simplex (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 2 | 2
Implant site abscess (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 9 | 3 | 12
Kidney infection (Infections and infestations) | 1 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1 | 1
Localised infection (Infections and infestations) | 2 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 8 | 1 | 9
Nail tinea (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 22 | 5 | 27
Oral candidiasis (Infections and infestations) | 1 | 0 | 1
Peritoneal infection (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 2 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 1
Postoperative infection (Infections and infestations) | 2 | 1 | 3
Prostate infection (Infections and infestations) | 1 | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 5 | 2 | 7
Skin infection (Infections and infestations) | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 4 | 0 | 4
Tooth infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 16 | 7 | 23
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 5 | 0 | 5
Viral infection (Infections and infestations) | 4 | 1 | 5
Viral upper respiratory tract infection (Infections and infestations) | 5 | 0 | 5
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0 | 2
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 5 | 4 | 9
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Electric shock (Injury, poisoning and procedural complications) | 1 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 7 | 2 | 9
Fall (Injury, poisoning and procedural complications) | 5 | 0 | 5
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 1 | 2
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 2
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 1 | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 1 | 3
Post procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural nausea (Injury, poisoning and procedural complications) | 4 | 0 | 4
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 2 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 8 | 4 | 12
Skin laceration (Injury, poisoning and procedural complications) | 2 | 1 | 3
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 2 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 2 | 2 | 4
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 2
Bacteria stool identified (Investigations) | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Blood bicarbonate decreased (Investigations) | 4 | 1 | 5
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Blood calcium decreased (Investigations) | 4 | 2 | 6
Blood chloride increased (Investigations) | 2 | 0 | 2
Blood cholesterol increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 6 | 1 | 7
Blood glucose increased (Investigations) | 2 | 0 | 2
Blood parathyroid hormone increased (Investigations) | 1 | 2 | 3
Blood phosphorus decreased (Investigations) | 1 | 1 | 2
Blood potassium decreased (Investigations) | 1 | 0 | 1
Blood potassium increased (Investigations) | 1 | 0 | 1
Blood pressure decreased (Investigations) | 1 | 2 | 3
Blood pressure increased (Investigations) | 9 | 4 | 13
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 1
Blood triglycerides increased (Investigations) | 2 | 0 | 2
Blood urea increased (Investigations) | 2 | 0 | 2
Blood uric acid increased (Investigations) | 1 | 2 | 3
Body temperature increased (Investigations) | 3 | 1 | 4
Cardiac murmur (Investigations) | 3 | 0 | 3
Cardiac stress test abnormal (Investigations) | 1 | 0 | 1
Culture positive (Investigations) | 0 | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 1 | 1
Electrocardiogram P wave abnormal (Investigations) | 1 | 0 | 1
Electrocardiogram PR shortened (Investigations) | 1 | 0 | 1
Electrocardiogram ST segment abnormal (Investigations) | 3 | 1 | 4
Electrocardiogram ST-T segment abnormal (Investigations) | 1 | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 1 | 0 | 1
Electrocardiogram abnormal (Investigations) | 1 | 0 | 1
Glucose urine present (Investigations) | 1 | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0 | 1
Haematology test abnormal (Investigations) | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 3 | 0 | 3
Heart rate decreased (Investigations) | 1 | 0 | 1
Heart rate increased (Investigations) | 3 | 1 | 4
Heart rate irregular (Investigations) | 2 | 0 | 2
International normalised ratio fluctuation (Investigations) | 1 | 0 | 1
International normalised ratio increased (Investigations) | 2 | 0 | 2
Liver function test abnormal (Investigations) | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 1
Platelet count increased (Investigations) | 1 | 0 | 1
Prostate examination abnormal (Investigations) | 0 | 1 | 1
Protein urine present (Investigations) | 1 | 0 | 1
Prothrombin time ratio increased (Investigations) | 1 | 0 | 1
Red blood cell count decreased (Investigations) | 2 | 0 | 2
Red blood cells urine positive (Investigations) | 1 | 0 | 1
Right ventricular systolic pressure increased (Investigations) | 1 | 0 | 1
Tandem gait test abnormal (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 1 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 3
Gout (Metabolism and nutrition disorders) | 3 | 1 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 2 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Oral intake reduced (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 6 | 15
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 2 | 18
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 2 | 10
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 1 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 7 | 21
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Epithelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 1
Burning sensation (Nervous system disorders) | 2 | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 2 | 0 | 2
Coordination abnormal (Nervous system disorders) | 2 | 0 | 2
Dizziness (Nervous system disorders) | 16 | 5 | 21
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Encephalomalacia (Nervous system disorders) | 1 | 0 | 1
Extensor plantar response (Nervous system disorders) | 0 | 1 | 1
Hand-arm vibration syndrome (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 16 | 10 | 26
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 1
Hyperreflexia (Nervous system disorders) | 1 | 2 | 3
Hypoaesthesia (Nervous system disorders) | 12 | 4 | 16
Hyporeflexia (Nervous system disorders) | 0 | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1
Lethargy (Nervous system disorders) | 3 | 1 | 4
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 19 | 3 | 22
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 2 | 0 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 2 | 1 | 3
Tremor (Nervous system disorders) | 4 | 0 | 4
Agitation (Psychiatric disorders) | 1 | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 4 | 1 | 5
Confusional state (Psychiatric disorders) | 1 | 2 | 3
Depressed mood (Psychiatric disorders) | 2 | 0 | 2
Depression (Psychiatric disorders) | 4 | 1 | 5
Emotional distress (Psychiatric disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 4 | 4 | 8
Major depression (Psychiatric disorders) | 0 | 1 | 1
Mood altered (Psychiatric disorders) | 1 | 0 | 1
Nervousness (Psychiatric disorders) | 1 | 1 | 2
Panic attack (Psychiatric disorders) | 2 | 0 | 2
Restlessness (Psychiatric disorders) | 0 | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 3 | 0 | 3
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Micturition disorder (Renal and urinary disorders) | 2 | 0 | 2
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 3 | 4
Renal failure chronic (Renal and urinary disorders) | 2 | 1 | 3
Renal impairment (Renal and urinary disorders) | 6 | 3 | 9
Urethral meatus stenosis (Renal and urinary disorders) | 1 | 0 | 1
Urethral stricture (Renal and urinary disorders) | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Breast discharge (Reproductive system and breast disorders) | 1 | 0 | 1
Breast discomfort (Reproductive system and breast disorders) | 1 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 1
Penile discharge (Reproductive system and breast disorders) | 1 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 1
Scrotal angiokeratoma (Reproductive system and breast disorders) | 1 | 0 | 1
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Bronchial hyperactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 8 | 28
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 5
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 3 | 14
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 4 | 17
Pleural rub (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 7
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 9
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 8
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Angiokeratoma (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Anhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 3 | 5
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 3 | 10
Pruritus allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 4 | 7
Vascular skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Arterial stenosis (Vascular disorders) | 1 | 0 | 1
Atherosclerosis (Vascular disorders) | 0 | 1 | 1
Flushing (Vascular disorders) | 2 | 2 | 4
Haematoma (Vascular disorders) | 1 | 0 | 1
Hot flush (Vascular disorders) | 2 | 1 | 3
Hypertension (Vascular disorders) | 5 | 2 | 7
Hypotension (Vascular disorders) | 3 | 1 | 4
Labile hypertension (Vascular disorders) | 1 | 0 | 1
Lymphoedema (Vascular disorders) | 2 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 1
Pallor (Vascular disorders) | 2 | 2 | 4
Peripheral coldness (Vascular disorders) | 2 | 1 | 3
Phlebitis (Vascular disorders) | 1 | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 1
Steal syndrome (Vascular disorders) | 1 | 0 | 1
Vascular pseudoaneurysm (Vascular disorders) | 1 | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0 | 1
Venous insufficiency (Vascular disorders) | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
No valid conclusions can be made from the predefined primary efficacy analysis. The sponsor believes that it is more statistically appropriate to compare placebo patients with Fabrazyme patients as they were randomized in the original Phase 4 trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, Principal Investigator (PI) can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.